CLINICAL TRIAL: NCT04404751
Title: Effectiveness of Quadruple Fortified Salt in Improving Hemoglobin Levels Among Anemic Women of Reproductive Age (18-49 Years) in Rural Low Resource Setting
Brief Title: Quadruple Fortified Salt Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydom Lutheran Hospital (Other)
Collaborators: University of Toronto (Other); Tanzania Food and Drugs Authority (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Salt_HGHRC#01
Record Dates: First submitted 2019-09-03; First posted 2020-05-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — iodized salt; Iron; Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Active Comparator)
  Interventions: Combination Product: Iodised salt with Iron, Folic acid and Vitamin B12
- Arm 2 (Active Comparator)
  Interventions: Combination Product: Iodised salt with Iron, Folic acid and Vitamin B12
- Arm 3 (Sham Comparator)
  Interventions: Combination Product: Iodised salt with Iron, Folic acid and Vitamin B12

INTERVENTIONS:
Combination Product: Iodised salt with Iron, Folic acid and Vitamin B12 — Fortified salt with either Iron and Iodine only or Fortified salt with Iodine, iron, Folic acid and Vitamin B12 compared with standard Iodized salt
  Other Names: Iodised salt with Iron

SUMMARY:
Anaemia is the world leading cause of disability and is responsible for about more than 115,000 maternal deaths and 591,000 perinatal deaths per year, of which 3/4 occur in Africa and Asia. Despite the fact that there are several causes of anemia, the most important causes are due to micronutrients deficiency, namely iron, Folic acid and Vitamin B12. Low intakes of these micronutrients consequently affect a woman's health, pregnancy outcome and the nutritional status of breast-fed children. With these in mind we wish to test the effectiveness of salt fortified with these four micronutrients (Iodine, Iron, Folic acid and vitamin B12) in raising the Hemoglobin levels among the non-pregnant and non-lactating women of reproductive age.

DETAILED DESCRIPTION:
Anaemia is the low level of Haemoglobin based on the location. As per WHO a woman is termed anaemic if has HB <11g/dl but in high attitude is =<13g/dl

ELIGIBILITY:
Inclusion Criteria:

* Adult with relative low haemoglobin (Hb level 8g/dl to 13g/dl)
* Able to eat food cooked with salt
* Able to give consent

Exclusion Criteria:

* Planning to become pregnant within the study period,
* chronically ill,
* have haematological diseases during study time,
* restricted to use salt in food

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Haemoglobin level | 10 months of consuming fortified salt
  After 10months use of quadruple fortified salt we expect the HB to rise by at least 50% as compared to those who used iodised salt

SECONDARY OUTCOMES:
Iron store replenishment | 10months of intervention
  The quadruple fortified salt is expected to replenish the iron store 100% after 10 months use of QFS

CONTACTS AND LOCATIONS:
Locations (1):
- Haydom Lutheran Hospital, Manyara, Tanzania